CLINICAL TRIAL: NCT04809168
Title: Prevalence of Spinal Neuropathic Pain in Ankylosing Spondylitis Patients and it's Impact on Sleep Quality: a Case-control Study
Brief Title: Neuropathic Spinal Pain in Ankylosing Spondylitis
Status: Active, not recruiting | Type: Observational
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Taciser Kaya, Associate professor, MD, Bozyaka Training and Research Hospital
Other Study IDs: 46418926TK
Record Dates: First submitted 2021-03-19; First posted 2021-03-22 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Surveys and Questionnaires; Equipment and Supplies; Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- AS patients: AS patients diagnosed according to the modified New York criteria
  Interventions: Other: Questionnaires and inventories
- Control: Age- and sex-matched control subjects with nociceptive/mechanical pain complaint lasting more than three months
  Interventions: Other: Questionnaires and inventories

INTERVENTIONS:
Other: Questionnaires and inventories — questionnaires and inventories related to primary end secondary outcomes will be applied and physical examination will be performed.
  Other Names: physical examination

SUMMARY:
The aim of this study is to investigate prevalence of neuropathic spinal pain in AS patients and it's impact on sleep quality. Moreover effects of neuropathic pain on quality of life and fatigue will be assessed.

DETAILED DESCRIPTION:
Ankylosing spondylitis (AS) is a chronic, inflammatory rheumatic disease that mainly presenting with chronic back pain. In general, chronic low back pain is currently defined as a mixed pain including nociceptive and neuropathic properties. Nociceptive pain in several rheumatic diseases displays neuropathic characteristics over time. Patients with AS are suffered from spinal, entheseal pain or pain originated from peripheral and root joints. Although being scarce, there are trials investigating and reporting neuropathic component of spinal pain in axial spondyloarthritis/ankylosing spondylitis patients. However these trials either are not controlled or did not specify painful region of interest. In a few controlled trials control subjects were not defined clearly.

Sleep problems are reported to be prevalent among patients with chronic pain conditions such as inflammatory rheumatic diseases and fibromyalgia. In patients with ankylosing spondylitis sleep disturbance is a well defined issue. The fact that sleep problem is a common problem in AS, raises the need to explore it's associates. In the trials measuring spinal neuropathic pain, sleep disturbances and it's association with neuropathic pain were not assessed.

So, investigators have aimed to investigate prevalence of neuropathic spinal pain in AS patients and it's impact on sleep quality. For this purpose a case-control study design was planned. Age- and sex-matched control subjects will be chosen among individuals submitted to out-patient clinic with nociceptive/mechanical pain complaint lasting more than three months. Participants in control group will be subjected to same exclusion criteria too.

This design will allow the investigators to determine whether spinal pain in AS patients displays neuropathic character more frequently than any chronic nociceptive pain does.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with AS according to the 1984 Modified New York Criteria
* Visual Analogue Scale (VAS) spinal pain score ≥ 2

Exclusion Criteria:

* Diabetes mellitus, renal insufficiency, hypothyroidism
* Carpal tunnel syndrome, postherpetic neuralgia, spinal cord compression
* Neurological diseases leading to neuropathic pain
* Cervical and lumbar radiculopathy
* Fibromyalgia
* Malignancy
* Severe cardiac disease
* Pregnancy
* Muscle weakness or hypoesthesia indicating peripheral nerve injury
* In the last three months medical treatment leading to neuropathy (colchicine etc.)
* In the last three months drug use for the treatment of fibromyalgia, depression and anxiety

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AS patients and age- and sex-matched control subjects will be chosen among individuals submitting to our out-patient clinic with nociceptive/mechanical pain complaint lasting more than three months.
Sampling Method: Non-Probability Sample
Enrollment: 292 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2024-11-02 (Actual); Study Completion 2025-12-02 (Estimated)

PRIMARY OUTCOMES:
Neuropathic pain | Once, at baseline
  It will be assessed using the PainDETECT questionnaire. This questionnaire contains nine questions all of which are self-report. Seven items are rated on a six point Likert scale and thus are scored between 0-5. These seven questions query some sensations such as burning, tingling or prickling, allodynia, numbness etc. Apart from these seven items, one item assesses the radiation of pain and the other one item looks for the temporal characteristics of pain. A total score of 12 or less indicates neuropathic component is unlikely, 13-18 means possible neuropathic component and 19 or greater means a neuropathic component is likely. Beside these, there are three items in a separate section measuring severity of pain at the time of evaluation, on average and maximum over the past month. This section is not taken into account in scoring
Sleep quality | Once, at baseline
  It will be assessed using Pittsburgh Sleep Quality Index (PSQI). It was developed by Buysse and coworkers in 1989. This index measures sleep quality quantitatively and covers 24 questions. Nineteen questions are self-rated and scoring is based on these self-rated questions, other five questions that rating by partner are not taken into account while calculating total score. Questionnaire measures seven domains; subjective sleep quality (question 6), sleep latency (question 2 and 5a), sleep duration (question 4), habitual sleep efficiency (question 1,3,4), sleep disturbances (question 5b-j), use of sleep medication (question 7), and daytime dysfunction (question 8 and 9) over the last month. Seven domain scores give a result on a 0 to 3 scale. To yield a total score the domain scores are summed. Total score varies between 0 and 21. Higher scores indicate worse sleep quality.

SECONDARY OUTCOMES:
Health related quality of life | Once, at baseline
  Health related quality of life will be assessed using (Ankylosing Spondylitis Quality of Life Questionnaire (ASQoL) querying symptoms, functioning, and disease-related concern. It covers 18 dichotomous questions that ask participants to answer in a yes or no fashion. An answer of "yes" is assumed as one point. To get a final score, all points are summed. Thus, total score is between 0-18 and higher scores indicate worse quality of life.
Fatigue | Once, at baseline
  It will be assessed using Fatigue Severity Scale. This scale contains nine questions and measures fatigue severity during the past week. Each question is rated between 1 (strongly disagree)-7 (strongly disagree). Total score is mean of all To calculate total score first the points of all answers are summed and then the result is divided by nine. Higher scores indicate severe fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Taciser Kaya, Study Director — Izmir Bozyaka Training and Reseach Hospital
Locations (1):
- Izmir Bozyaka Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aydin E, Bayraktar K, Turan Y, Omurlu I, Tastaban E, Sendur OF. [Sleep quality in patients with ankylosing spondylitis]. Rev Bras Reumatol. 2015 Jul-Aug;55(4):340-5. doi: 10.1016/j.rbr.2014.12.007. Epub 2015 Feb 9. Portuguese. PMID 25772656
- [Background] Geler-Kulcu D, Batibay S, Ozturk G, Mesci N. The association of neuropathic pain and disease activity, functional level, and quality of life in patients with ankylosing spondylitis: a cross-sectional study. Turk J Med Sci. 2018 Apr 30;48(2):257-265. doi: 10.3906/sag-1707-147. PMID 29714437
- [Background] Choi JH, Lee SH, Kim HR, Lee KA. Association of neuropathic-like pain characteristics with clinical and radiographic features in patients with ankylosing spondylitis. Clin Rheumatol. 2018 Nov;37(11):3077-3086. doi: 10.1007/s10067-018-4125-z. Epub 2018 Apr 30. PMID 29713968
- [Background] Wu Q, Inman RD, Davis KD. Neuropathic pain in ankylosing spondylitis: a psychophysics and brain imaging study. Arthritis Rheum. 2013 Jun;65(6):1494-503. doi: 10.1002/art.37920. PMID 23460087
- [Background] Li Y, Zhang S, Zhu J, Du X, Huang F. Sleep disturbances are associated with increased pain, disease activity, depression, and anxiety in ankylosing spondylitis: a case-control study. Arthritis Res Ther. 2012 Oct 11;14(5):R215. doi: 10.1186/ar4054. PMID 23058191